CLINICAL TRIAL: NCT04517734
Title: Erythroferrone and Its Impact on Maternal and Neonatal Iron Homeostasis
Status: Completed | Type: Observational
Sponsor: Cornell University (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: 0911001050
Record Dates: First submitted 2020-08-11; First posted 2020-08-18 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Pregnancy Anemia; Newborn; Anemia
MeSH Terms: conditions — Anemia, Neonatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During pregnancy 15 mL maternal blood sample collected. At delivery 15 mL maternal blood sample, 20 mL umbilical cord blood sample and the placenta are collected.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant Adolescents
- Pregnant Women Carrying Multiple Fetuses

SUMMARY:
Erythroferrone (ERFE) is a recently identified iron-regulatory hormone that couples iron homeostasis to erythropoiesis but at this time there are no human data on this hormone in pregnant women and their neonates. The investigators hypothesize that ERFE is a sensitive biomarker of iron deficiency and anemia in pregnancy and neonates, and that it mediates the feedback mechanism to correct iron deficiency and anemia. To address this research gap, the investigators will measure ERFE in maternal serum, umbilical cord serum and placental tissue using an existing biospecimen archive.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant volunteers

Exclusion Criteria:

* Hemoglobinopathies
* Pre-existing diabetes
* Malabsorption diseases
* Pregnancy induced hypertension
* Elevated diastolic blood pressure (>110)
* Previous treatment for lead exposure or elevated childhood lead concentrations.
* Preexisting medical conditions known to impact iron homeostasis

Ages: 11 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant women carrying multiple fetuses (twins, triplets and quadruplets) or pregnant adolescents carrying a single fetus
Sampling Method: Non-Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Maternal Erythroferrone During Pregnancy | Measures will be obtained from maternal blood collected throughout the 40 weeks of pregnancy
Maternal Erythroferrone at Delivery | Measures will be obtained from maternal blood collected at delivery
Neonatal Erythroferrone at Birth | Measures will be obtained from umbilical cord blood collected at delivery
Placental Erythroferrone mRNA and Ferroportin protein Expression | Measures will be obtained from placental samples collected at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly O'Brien, PhD, Principal Investigator — Cornell University; Elizabeta Nemeth, PhD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Rochester Adolescent Maternity Program, Rochester, New York
  - Strong Memorial Hospital, Rochester, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Delaney KM, Guillet R, Pressman EK, Ganz T, Nemeth E, O'Brien KO. Serum Erythroferrone During Pregnancy Is Related to Erythropoietin but Does Not Predict the Risk of Anemia. J Nutr. 2021 Jul 1;151(7):1824-1833. doi: 10.1093/jn/nxab093. PMID 33982118